CLINICAL TRIAL: NCT07336212
Title: Impact of Restorative Treatment on Occlusal Characteristics and Masseter Muscle Activity in Children With Molar-Incisor Hypomineralization: A T-Scan and sEMG Pilot Study
Brief Title: Impact of Glass-Hybrid Restoration on Occlusal Force Distribution and Masticatory Muscle Activity in Children With Molar-Incisor Hypomineralization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pedo-occlusion
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Molar-Incisor Hypomineralization (MIH)
Keywords: Pediatric Dentistry; MIH; Occlusal Balance; Electromyography; T-Scan; sEMG; Molar-Incisor Hypomineralization; Occlusal Force Distribution; Glass-Hybrid Restoration
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glass-Hybrid Restoration in MIH-Affected Molars (Experimental): Participants receive restorative treatment of symptomatic, carious first permanent molars affected by molar-incisor hypomineralization using a bulk-fill glass-hybrid restorative material (Equia Forte®). Functional assessments, including digital occlusal analysis with the T-Scan system and surface electromyography (sEMG) recordings of the masseter and anterior temporalis muscles, are performed at baseline and 3 months after restoration.
  Interventions: Procedure: Glass-Hybrid Restoration

INTERVENTIONS:
Procedure: Glass-Hybrid Restoration — Selective caries removal followed by bulk-fill glass-hybrid restoration of MIH-affected first permanent molars using Equia Forte®. The procedure is performed by a calibrated pediatric dentist according to the manufacturer's instructions. Occlusion is checked and adjusted after restoration prior to functional assessments.

SUMMARY:
This prospective pilot study evaluates the effect of restoring symptomatic, carious molar-incisor hypomineralization (MIH)-affected permanent molars using a glass-hybrid restorative material on occlusal force distribution and masticatory muscle activity. Digital occlusal analysis using the T-Scan system and surface electromyography (sEMG) recordings of the masseter and anterior temporalis muscles are performed before treatment and three months after restoration. Hypersensitivity is assessed using the Schiff Cold Air Sensitivity Scale.

DETAILED DESCRIPTION:
This single-arm prospective pilot study investigates whether restorative rehabilitation of MIH-affected permanent molars leads to functional improvements in occlusal balance and neuromuscular activity. Children aged 7-13 years with symptomatic MIH requiring restorative treatment undergo standardized glass-hybrid restorations. Functional occlusal analysis is conducted using the T-Scan Novus system to assess lateral occlusal force distribution, while bilateral surface electromyography (sEMG) evaluates masseter and temporalis muscle activity during maximum voluntary clenching. Dentin hypersensitivity is assessed using the Schiff Cold Air Sensitivity Scale. Pre- and post-treatment outcomes are compared to explore early functional adaptation following MIH rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7 to 13 years
* Diagnosis of molar-incisor hypomineralization (MIH) according to the criteria of Ghanim et al.
* Presence of at least two MIH-affected first permanent molars with post-eruptive enamel breakdown requiring restorative treatment
* Presence of dentin hypersensitivity in the affected molars
* Ability to comply with T-Scan and surface electromyography (sEMG) recording procedures
* Written informed consent obtained from parents or legal guardians, and assent from the child
* Exclusion Criteria:
* Previous or ongoing orthodontic treatment
* Presence of craniofacial anomalies or syndromes
* Diagnosis of temporomandibular disorders
* Parafunctional habits (e.g., bruxism)
* Clinically evident facial asymmetry
* Malocclusions such as crossbite or open bite
* Systemic diseases or medications affecting neuromuscular function -Inability to cooperate with functional assessment procedures -

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Lateral Occlusal Force Distribution (LOFD) | Baseline and 3 months post-treatment
  Change in lateral occlusal force distribution assessed using the T-Scan digital occlusal analysis system during maximum voluntary clenching. The primary variable is the absolute deviation from ideal 50-50 bilateral force distribution, calculated at baseline and 3 months after glass-hybrid restoration.

SECONDARY OUTCOMES:
Masticatory Muscle Activity Symmetry | Baseline and 3 months post-treatment
  right-left asymmetry indices of the masseter and anterior temporalis muscles measured using surface electromyography (sEMG) during maximum voluntary clenching.
Dentin Hypersensitivity | Baseline and 3 months post-treatment
  Dentin hypersensitivity of MIH-affected molars assessed using the Schiff Cold Air Sensitivity Scale following an air-blast stimulus.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No